CLINICAL TRIAL: NCT01278004
Title: A Randomised Double-blind Placebo-controlled Trial of the Safety and Efficacy of Ethosuximide 250mg Capsules for the Management of Chemotherapy Induced Painful Peripheral Neuropathy
Brief Title: Chemotherapy Induced Painful Peripheral Neuropathy Ethosuximide (The CIN-E Study)
Acronym: CINE-E
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CCR3116
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Cancer; Peripheral Neuropathy
Keywords: Adult cancer patients with chemotherapy-induced painful peripheral neuropathy
MeSH Terms: conditions — Neoplasms; Peripheral Nervous System Diseases | interventions — Ethosuximide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Drug: Placebo
- Drug (Experimental)
  Interventions: Drug: Ethosuximide

INTERVENTIONS:
Drug: Ethosuximide — Drug will be dose escalated in order to reach maximum tolerated dose starting with 250mg.
  Arms: Drug
Drug: Placebo — Capsule
  Arms: Placebo

SUMMARY:
This study is a drug trial of ethosuximide as a painkiller if you develop pain as a side effect of chemotherapy. Ethosuximide will be compared against placebo (an inactive substance) to test whether any response is a true effect of the drug, and not a 'placebo effect'.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18
* Diagnosis of cancer
* Willing and able to give informed consent to the CIN-E study and complete study questionnaires, this involves adequate understanding of written and spoken English (translators will not be used)
* Chemotherapy-induced painful peripheral neuropathy as diagnosed by score of >12 on the Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) with a pain intensity rating of >4, on a 11 point numeric rating scale (0= no pain, 10= worst possible pain).
* Duration of chemotherapy-induced painful peripheral neuropathy >4 weeks. Participant may either have completed chemotherapy, or be receiving ongoing chemotherapy.
* Able to attend research centre according to the required visit schedule.
* Diet allows bovine gelatine (present in both ethosuximide and placebo capsules)
* Women of child-bearing potential must be using a reliable form of contraception i.e. oral contraceptives, a barrier method (condom or diaphragm), intra-uterine device or abstinence.

Exclusion Criteria:

* Renal impairment (serum creatinine >1.5x normal level)
* Deranged liver function (AST>3x normal level)
* Patients currently taking any anti-depressant medication, for example fluoxetine, paroxetine, citalopram, venlafaxine, amitriptyline, or within the past week.
* Patients currently taking any other anti-epileptic drug, including gabapentin, or within the past week.
* Pregnancy
* Allergy to succinimides, ethosuximide, methsuximide, phensuximide. Pre-exisitng painful peripheral neuropathy of any other cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Reduction in pain intensity from baseline to endpoint as assessed on a Numerical Pain Rating scale. | 6 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - The Royal Marsden NHS Foundation Trust, London